CLINICAL TRIAL: NCT00678977
Title: A Phase I, Open-label, Study of the Safety, Tolerability and Pharmacokinetics of Pazopanib in Combination With Gemcitabine and Gemcitabine Plus Cisplatin for Advanced Solid Tumors
Brief Title: A Phase I, Open-label, Study of Pazopanib in Combination With Gemcitabine and Gemcitabine Plus Cisplatin for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG109599
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: pharmacokinetics; cisplatin; pazopanib (GW786034); Solid tumors; anti-angiogenesis; gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Dose Escalation - Patients will be entered into dose cohorts of three patients. Each cohort will be assigned to a dose level for the duration of the study. There will be no intra-patient dose-escalation. The starting dose will be 400 mg daily of pazopanib, and 1000 mg/m2 gemcitabine. Intermediate dose levels may also be explored. Intravenous gemcitabine will be given on Day 1 and 8 of Cycle 1 and each subsequent cycle.
  Cohort expansion phase - patients will receive gemcitabine alone, at the OTR dose starting on Day 1 of Cycle 1. Pazopanib will be administered at the OTR beginning on Day 2 Cycle 1 after the last blood sample for gemcitabine analysis is collected, and pazopanib administration will continue for the duration of the study. Patients will return to the clinic on Day 8 of Cycle 1 for simultaneous administration of gemcitabine and pazopanib. On Day 1 of Cycle 2 patients will receive the simultaneous administration of gemcitabine and pazopanib
  Interventions: Drug: Pazopanib (GW786034); Drug: Gemcitabine
- Arm B (Experimental): Dose Escalation - Patients will be entered into dose cohorts of three patients. Each cohort will be assigned to a dose level for the duration of the study. There will be no intra-patient dose-escalation. The starting dose will be 400 mg daily of pazopanib, 1000 mg/m2 gemcitabine and 60 mg/m2 cisplatin. Doses of gemcitabine may range from 600 to 1250 mg/m2. Doses of cisplatin may range from 60 to 80 mg/m2. Intermediate dose levels may also be explored. Pazopanib administered starting on Day 1 of Cycle 1, gemcitabine co-administration on Day 1 and 8, and cisplatin on Day 1 in each 21-day cycle.
  Cohort expansion - patients will receive gemcitabine and cisplatin alone, at the OTR doses, starting on Day 1 of Cycle 1. Pazopanib will be administered at the OTR dose beginning on Day 2 of Cycle 1, and pazopanib administration will continue for the duration of the study. Patients will return to the clinic on Day 8 of Cycle 1 for simultaneous administration of gemcitabine and pazopanib
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pazopanib (GW786034) — initial dose 400mg daily in 21-day cycles; increase in dose up to 800mg daily following evaluation of safety and tolerability
  Arms: Arm A
Drug: Gemcitabine — Gemcitabine on Days 1 and 8 of each cycle; initial dose 600 mg/m2 increase to 1,000mg/m2 after evaluation of safety and tolerability; increase to 1250mg/m2 after evaluation of safety and tolerability
Drug: Cisplatin — Cisplatin on Day 1 of each 21-day cycle initial dose 60mg/m2; increase to 80mg/m2 after evaluation of safety and tolerability
  Arms: Arm B

SUMMARY:
This is an open-label, two-arm, Phase I, dose escalation study to evaluate the safety and tolerability and to determine the optimal tolerated regimen(OTR) of pazopanib in combination with gemcitabine (Arm A) or pazopanib, gemcitabine, and cisplatin (Arm B) in patients with advanced solid tumors. Patients will be enrolled in cohorts of 3 to receive escalating doses of pazopanib and gemcitabine or pazopanib, gemcitabine and cisplatin. Dose escalation schemas for each study arm are described in the protocol. For each arm, the OTR will be defined as the highest dose combination of the agents where no more than one out of six patients experiences a dose-limiting toxicity. Six to twelve additional patients in each arm will be studied with the OTR to evaluate toxicity and pharmacokinetics. This will allow an assessment of potential drug-drug interactions. Antitumor activity will be assessed using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a histologically or cytologically confirmed advanced solid tumor, having failed standard therapy or for whom there is no standard therapy. Patients should have unresectable or metastatic disease.
* Age greater than or equal to 18 years
* Performance status must be ECOG 0-1.
* Prior therapies allowed: unlimited.
* Adequate organ function
* Patients must have measurable or evaluable disease:
* No unstable or serious concurrent condition.
* A female subject is eligible to enter and participate in the study if she is: Of non-childbearing potential
* Subjects must discontinue HRT prior to study enrolment due to the inhibition of CYP enzymes that metabolize estrogens and progestins.
* Childbearing potential, includes any female who has had a negative serum pregnancy test at screening and within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception.
* A male with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception or abstinence during the study.
* Patients must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up
* At least 4 weeks must have elapsed since last administration of chemotherapy and subjects must have recovered from any toxicity attributed to the agent prior to enrolment in this study.
* Prior radiotherapy is permissible, provided at least 4 weeks have elapsed since the last treatment to allow for full bone marrow recovery.
* Patients with metastatic disease to the brain should have definitive therapy for their brain metastases, should be asymptomatic. (Patients with previously treated brain metastases who are asymptomatic, off steroids and anti-seizure medications for greater than 3 months are eligible for study.)

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti seizure medication for one week prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required.
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480 msecs.
* History of any one of more of the following cardiovascular conditions within the past 6 months:

Cardiac angioplasty or stenting; myocardial infarction; unstable angina; symptomatic peripheral vascular disease; Class III or IV congestive heart failure as defined by the New York Heart Association

* Has had any major surgery, chemotherapy, investigational agent, biological therapy or hormonal therapy within the last 28 days and/or not recovered from a prior therapy.
* Any unstable or serious concurrent condition (e.g., active infection requiring systemic therapy)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of greater than or equal to 140mmHg or diastolic blood pressure (DBP) of greater than or equal to 90mmHg].
* History of cerebrovascular accident (CVA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Hemoptysis within 6 weeks prior to first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent, or compliance to study procedures.
* Is unable or unwilling to discontinue prohibited medications, as listed in Section 8.2 for 14 days or five half-lives of a drug prior to Visit 1 and for the duration of the study.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Prior use of an investigational or licensed tyrosine kinase inhibitor that targets VEGF receptors.

Note: Prior use of bevacizumab is allowed.

* Is now undergoing and/or has undergone in the 14 days immediately prior to first dose of study drug, any cancer therapy (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy).

Note: For prior bevacizumab therapy at least 40 days should have elapsed since last dose.

* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib, gemcitabine, or cisplatin. (To date there are no known FDA approved drugs chemically related to pazopanib).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04-03 (Actual); Primary Completion 2010-03-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Optimum tolerated regimen (OTR) for each regimen in each arm of the study. OTR determined evaluation of AEs and change in lab values. OTR defined as the highest dosing regimen that results in dose limiting toxicity in no more than 1 of 6 subjects | Until disease progression

SECONDARY OUTCOMES:
Anti-tumor activity evaluated using RECIST criteria (if subjects have measurable disease). Assessments of disease every 6 to 12 weeks, recorded as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD). | Until Disease progression
Pharmacokinetic parameters AUC(0-24), Cmax, and tmax of pazopanib, gemcitabine, and ultrafilterable platinum. | Dose Expansion - Cycle; Dose-Expansion Cycle 2
Levels of circulating cytokine and angiogenic factors (CAF) biomarkers (such as IL 2, IL-10, VEGF, sVEGFR2) in plasma will be determined | Day 1 of each cycle until disease progression
Genetic variants in select candidate genes in the host DNA will be evaluated | Day 1 of first cycle

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Essen, North Rhine-Westphalia, Germany
- GSK Investigational Site, Newcastle upon Tyne, Northumberland, United Kingdom

REFERENCES:
- [Background] Plummer R, Madi A, Jeffels M, Richly H, Nokay B, Rubin S, Ball HA, Weller S, Botbyl J, Gibson DM, Scheulen ME. A Phase I study of pazopanib in combination with gemcitabine in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2013 Jan;71(1):93-101. doi: 10.1007/s00280-012-1982-z. Epub 2012 Oct 11. PMID 23064954
- See also: Results for study VEG109599 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG109599?search=study&study_ids=VEG109599#rs